CLINICAL TRIAL: NCT04945850
Title: Can COVID-19 Persist in Intraocular Fluid?
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Sapna Gangaputra, Principal Investigator, Vanderbilt University Medical Center
Other Study IDs: 100800
Record Dates: First submitted 2021-06-17; First posted 2021-06-30 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Ocular Infection, Viral
MeSH Terms: conditions — Eye Infections, Viral

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Covid negative: 20 patients undergoing ocular surgery who are COVID negative will be included as control patients and undergo the same procedures.
  All patients will get a vitreous tap from operative eye 0.1-0.2 ml fluid. This fresh sample will be tubed to the lab using a unique marked label. This will be performed after the trocar is placed
  At the end of surgery, the BSS bag will be tubed to the lab using the same label.
  Interventions: Procedure: routine care intraocular sx
- Covid positive: 60 patients undergoing ocular surgery with previous COVID infection will be stratified into three groups by time since diagnoses: 3, 6, 12 months ~ 20 patients per group.
  All patients will get a vitreous tap from operative eye 0.1-0.2 ml fluid. This fresh sample will be tubed to the lab using a unique marked label. This will be performed after the trocar is placed
  At the end of surgery, the BSS bag will be tubed to the lab using the same label.
  Interventions: Procedure: routine care intraocular sx

INTERVENTIONS:
Procedure: routine care intraocular sx — Fluid was collected during routine intraocular surgery

SUMMARY:
Several common viruses thrive and persist in intraocular fluid due to ocular immune privilege. Immune privilege is maintained by lack of lymphatic tissue, a strong blood ocular barrier, and regulation of the systemic immune response via immunosuppressive factors such as TGF-B and processes like anterior chamber associated immune deviation. Notable viruses that benefit from ocular immune sequestration include DNA viruses such as Herpes simplex virus, Varicella Zoster, Cytomegalovirus and RNA viruses like Ebola and Rubella.In light of the global 2019 Severe acute respiratory syndrome coronavirus-2 virus (SARS CoV-2 or commonly COVID-19) pandemic, there has been growing interest on COVID-19's long term effects on the ocular system. Ocular symptoms at the time of diagnosis and during illness have been reported previously. The most commonly reported are epiphora, chemosis, and conjunctivitis. Less common were findings of retinal hemorrhages and retinal ischemic changes. Recent literature has demonstrated its presence in ocular fluid such as tears and the aqueous humor, but whether this is sustained for an extended period of time has yet to be determined. Long term effects of covid on the neurological system are being identified - large vessel ischemic strokes, cerebral hemorrhages, cranial nerve palsies, and memory loss in young adults are being reported. The persistence of COVID 19 in the intraocular fluid several months after covid infection has not been studied previously.

DETAILED DESCRIPTION:
Animal Studies and Previous Human Studies

Other coronavirus murine and feline models have shown ocular involvement. In Robbins et al experiment, mice underwent intracameral and intravitreal injections with murine coronavirus. Within 3 days, those with injections into the AC demonstrated a variety of findings such as keratitis and anterior uveitis; whereas those who underwent intravitreal injection had multilayered retinal lesions with RPE scarring and retinal atrophy. CNS disease and/or death occurred in a third of those from intravitreal injections. Viral antigens have been isolated from these mice but there is evidence immune cells and pro-inflammatory factors also contribute to the retinopathy findings. This murine model, known as Experimental CoV Retinopathy, has been used to examine host immune response that lead to retinal damage. Cats infected with feline infectious peritonitis virus, a feline coronavirus, manifested with conjunctivitis, pyogranulomatous anterior uveitis, retinal vasculitis, choroiditis and retinal detachment. Over 90% of the cats had antigen detected in the conjunctiva.

Viruses such as VZV, HSV, and CMV and parasites like Toxoplasmosis have been isolated from the intraocular fluid of human eyes using polymerase chain reaction (PCR), despite having normal or negative serum titers.

Enrollment/Randomization

Those who meet inclusion criteria will be provided an opportunity to participate in study. They will provide written informed consent in accordance with the HIPAA regulations and Vanderbilt IRB approval.

Study Procedures

* Patients selected for study:

  80 total patients

  20 patients undergoing ocular surgery who are COVID negative will be included as control patients and undergo the same procedures 60 patients undergoing ocular surgery with previous COVID infection will be stratified into three groups by time since diagnoses: 3, 6, 12 months ~ 20 patients per group.
  * All patients will get a vitreous tap from operative eye 0.1-0.2 ml fluid. This fresh sample will be tubed to the lab using a unique marked label. This will be performed after the trocar is placed
  * At the end of surgery, the BSS bag will be tubed to the lab using the same label.
* Informed consent will be obtained during pre-operative clinic visit
* Samples will get a special-colored label and tubed to Dr Schmitz and Dr. Maris lab from the OR

Laboratory analyses

VUMC MIDL Lab Testing Protocol:

• Specimens: 100-200ul dry taps of vitreous fluid will be delivered to the VUMC MIDL lab and frozen (-80C) until nucleic acid is extracted. 1L bags of BSS saline containing ocular fluid will be delivered to the VUMC MIDL lab and aliquoted into 3 10ml falcon tubes and then frozen (-80C) until nucleic acid is extracted.

Nucleic acid extraction:

• Specimens will have total RNA & DNA extracted on the easyMAG, EMAG, or EZ1 automated nucleic acid extraction platforms.

Real time RT-PCR:

• RNA present in nucleic acid extracts will be reverse transcribed into cDNA. Target cDNA will be amplified by PCR and target fluorescence emission will be measured and detected in real time. Targets include the N1 & N2 regions of the nucleocapsid gene of SARS-CoV-2, and an internal control to monitor for adequate nucleic acid extraction and absence of PCR inhibitors: human RNase P (RP). Target Ct values will be recorded from detected samples.

Next Generation Sequencing (NGS):

* Illumina: Nucleic acid extracts will undergo targeted SARS-CoV-2 whole genome amplification by tiling PCR. Amplicons will undergo DNA library preparation, barcoding, and QC. DNA libraries will be inoculated onto MiSeq flow cells and sequenced. Reads will be outputted as FASTQ files.
* MinION: Total nucleic acid extracts will undergo DNA library preparation, barcoding, and QC. DNA libraries will be inoculated onto MinION Mk1C & Flongle flow cells for metagenomic deep sequencing. Reads and associated quality data will be outputted as FASTQ files.

Risks

The study procedures involve minimal risk as they are performed in an eye that is undergoing an elective scheduled operative procedure for medical reasons. The safe and sterile procedure greatly decreases the risk.

Reporting of Adverse Events or Unanticipated Problems involving Risk to Participants or Others

Any adverse events will be reported to the Vanderbilt Eye Institute, and VUMC IRB per policy and procedure. These will be submitted within one week of occurrence.

Study Withdrawal/Discontinuation

VUMC IRB will be notified of study withdrawal and discontinuation. We anticipate the study to last approximately 1 year.

Data analysis:

Ct values from RT-PCR detected samples will be compared and correlated with clinical data. SARS-CoV-2 sequences from Illumina and MinION NGS platforms will be analyzed for variants and correlated with clinical data. non-SARS-CoV-2 microbial sequences will be analyzed and identified to the microbial species level. The ocular fluid 'microbiome' will be compared across samples and correlated with clinical data.

Privacy/Confidentiality Issues

Patient information will be de-identified and uploaded to REDCAP survey to ensure confidentiality and privacy.

Follow-up and Record Retention

The duration is expected to be one year. The data will be retained for six months following closure of the study. This will be destroyed afterward.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Proof of previous COVID-19 infection
* Patients scheduled for elective ocular surgery at Vanderbilt Medical Center

Exclusion Criteria:

• 17 years of age and younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We plan to recruit 80 patients to be enrolled in the study. This will be 20 COVID negative patients and 60 COVID positive patients stratified into three groups (20 per group) based on time since diagnosis as detailed above. This will provide sufficient sample size to be able to identify if the presence of covid in the eye is associated with prior infection and how long the virus can subsist in intraocular fluid.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-06-16 (Actual); Study Completion 2022-06-16 (Actual)

PRIMARY OUTCOMES:
Presence of Covid-19 | 12 months
  We aim to examine the presence of COVID-19 in the intraocular fluid.
Duration of persistent virus isolation | 12 months
  Duration of persistent virus isolation from intraocular fluid
Microbiological methods | 12 months
  microbiological methods of diagnosing.
Analyzing COVID-19 | 12 months
  Analyzing COVID-19 using ocular fluids.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
there is no specimen left